CLINICAL TRIAL: NCT05284682
Title: Metabolic Characterization of Patients With Dilated Cardiomyopathy a Prospective Case-control Study
Brief Title: Metabolic Characterization of Patients With Dilated Cardiomyopathy
Acronym: MECHAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MECHAD
Record Dates: First submitted 2021-11-19; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: DCM - Dilated Cardiomyopathy; Heart Failure
Keywords: Energy metabolism
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dilated cardiomyopathy: Patients with heart failure on the basis of dilated cardiomyopathy.
  Interventions: Diagnostic Test: Right hearted catheterization
- Control group without heart failure: Control group from the ablation laboratory without heart failure
  Interventions: Diagnostic Test: Right hearted catheterization

INTERVENTIONS:
Diagnostic Test: Right hearted catheterization — Right hearted catheterization and collection of blood sampels in the coronary sinus, arterial blood and central venous blood for analysis of energy substrate metabolites.

SUMMARY:
The overall aim of the study is to explore the energy metabolism of the failing heart.

Primary objective is to understand the differences in the energy metabolism in patients with DCM and heart failure compared to matched controls without heart failure. Secondary objectives, is to understand if optimal medical therapy, including sodium-gucose transporter 2 inhibitors (SGLT2i), alter the cardiac metabolism in DCM-patients. The investigators will also examine if changes in cardiac metabolism happens during exercise in patients with DCM.

This will be done with invasive measurements of a range of energy substrate metabolites in the coronary sinus of the heart in patients with heart failure due to DCM and controls without heart failure respectively. A range of other clinical characteristics will also be examined to characterize patients and controls.

DETAILED DESCRIPTION:
Study Design:

The MECHAD study is an explorative prospective cohort study with matched controls including patients with heart failure with reduced ejection fraction (HFrEF, EF≤40%) due to DCM in NYHA-class II-IV, ≥18 years, referred to Department of Cardiology/Sahlgrenska for heart failure work-up. A control group will be collected with age, gender and body mass index (BMI) matched controls without heart failure from the electrophysiology laboratory.

Study Site:

Sahlgrenska University Hospital is a tertiary center for patients in the need of heart failure evaluation, staging and therapy. Further, Sahlgrenska University Hospital is included in the assignment as one of the national centers for heart transplantation in Sweden. Patients with advanced HF are referred from the western and northern parts of Sweden and as part of clinical evaluation they most often undergo transthoracic echocardiogram (TTE), cardiopulmonary exercise test (CPET) as well as right-sided heart catheterization (RHC) with biopsy from the right ventricle septum or the lateral wall in the left ventricle. The site receives approximately 150 patients for evaluation every year and about 70% have clinically DCM.

Patient information and consent:

The Principal Investigator (or delegated sub investigator) will provide each patient with verbal and written information regarding the objectives and procedures of the study and possible risks involved. The patients will be informed about their right to withdraw from the study at any time. Prior to any study related procedures, the informed consent will be reviewed, signed and dated by the patient and investigator. The research unit at the Department of Cardiology/Sahlgrenska University hospital have dedicated research nurses who will facilitate coordination of the study.

Study timetable:

The inclusion in the study is planned to start in Q1 2022 and will continue until 30 patients with HF and 60 patients without HF (controls) are included. The investigators estimate to be able to include one patient per week in average.

Power Calculation and statistical analyses The investigators aim to include 30 patients with HF and 60 matched patients without HF as controls. To calculate the power, data was used from one study in humans showing an increase in 3-hydroxybutanoyl from 0.29 pmol/mg in a non-failing heart to 0.59 pmol/mg in failing heart. This large difference would result in only 2 patients in each group. However, the estimated increase in 3-hydroxybutanoyl does not directly transmitted to our cohort of DCM, therefore a larger sample was chosen.

ELIGIBILITY:
For cases (Heart Failure on the basis of DCM)

Inclusion Criteria:

* Signed and dated the Informed Consent Form
* Male and female subjects ≥18 years of age
* Chronic Heart failure (HF) with LVEF ≤40%
* HF due to dilated cardiomyopathy (DCM)
* New York Heart Association (NYHA) class ≥2
* Treatment with basic optimal medical therapy.
* Clinical indication for invasive evaluation of heart failure

Exclusion Criteria:

* Life expectancy < 3 years due to other reasons than cardiovascular, cardiac transplantation or left ventricular assist device
* Diabetes mellitus type 1 and 2
* Known hereditary hypercholesterolemia
* Ongoing lipid lowering therapy
* Patients on ketogenic diets
* BMI>35 or <19
* Pregnancy
* Any current life-threatening cardiac dysrhythmia, cardiac surgery, acute coronary syndrome, or non-elective percutaneous coronary intervention (PCI) <3 months
* Current significant major or unstable respiratory disease
* Considerable hematological disease, hepatic disease, renal disease and/or gastrointestinal disease
* Stroke, transient ischemic attack, carotid surgery or angioplasty <3months
* estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI formula) <30 mL/min/1.73m2 or patients on renal dialysis
* Expected inability (by the investigator) to comply with the protocol
* Subjects incapable to giving consent personally

For control subjects (no heart failure)

Inclusion criteria:

* Signed and dated Informed Consent Form
* Male and female subjects ≥18 years of age
* Clinical indication for electrophysiology examination

Exclusion criteria:

* Heart Failure (HFpEF, heart failure with mid-range ejection fraction (HFmrEF) or HFrEF)
* Life expectancy < 3 years due to other reasons than cardiovascular, cardiac transplantation or left ventricular assist device
* Diabetes mellitus type 1 and 2
* Known hereditary hypercholesterolemia
* Ongoing lipid lowering therapy
* Patients on ketogenic diets
* BMI>35 or <19
* Pregnancy
* Any current life-threatening cardiac dysrhythmia, cardiac surgery, acute coronary syndrome, or non-elective PCI <3 months
* Current significant major or unstable respiratory disease
* Considerable hematological disease, hepatic disease, renal disease and/or gastrointestinal disease
* Stroke, transient ischemic attack, carotid surgery or angioplasty <3months,
* eGFR by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI formula) <30 mL/min/1.73m2 or patients on renal dialysis
* Expected inability (by the investigator) to comply with the protocol
* Subjects incapable to giving consent personally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sahlgrenska University Hospital is a tertiary center for patients in the need of heart failure evaluation. Further, Sahlgrenska University Hospital is included in the assignment as one of the national centers for heart transplantation in Sweden. Patients with advanced HF are referred from the western and northern part of Sweden and as part of clinical evaluation they most often undergo transthoracic echocardiogram (TTE), cardiopulmonary exercise test (CPET) and right-sided heart catheterization (RHC) with myocardial biopsy. The site receives approximately 150 patients for evaluation every year and about 70% have clinically DCM. The study population will be will be recruited from this population.
  The control population of the study will be recruited from the electrophysiology laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic markers | through study completion, on average 2 years
  Energy substrate metabolic markers in arterial blood and coronary sinus for the calculation of energy metabolism in the myocardium.

SECONDARY OUTCOMES:
Metabolic markers after medical optimization | through study completion, on average 4 years
  Energy substrate metabolic markers in arterial blood and coronary sinus for the calculation of energy metabolism in the myocardium.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Ljungman, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Western Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No